CLINICAL TRIAL: NCT02160028
Title: Pain and Placebo Analgesia. A Double Blinded, Randomized, Clinical Study About the Impact of Information About Anesthesia, and the Experience of Pain and Stress During Dental Treatment.
Brief Title: Pain and Placebo Analgesia. Does Extended Information About Dental Procedures Reduce Pain Induced by Dental Treatment?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Bergen (Other); Tannhelsetjenestens Kompetansesenter Vest, TK Vest (Unknown); Tannlegesenteret Madlagården, TSMG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014/2615/SGK
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Anxiety; Odontophobia
Keywords: Information; Pain; Stress; Fear; Placebo analgesia
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Anesthetics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard information (Active Comparator): This group is given anesthetics and standard information before dental treatment about the anesthetics.
  Interventions: Other: anesthetics and standard information before dental treatment
- Extended information (Experimental): This group is given anesthetics and extended information before dental treatment about the anesthetics.
  Interventions: Other: anesthetics and extended information before dental treatment

INTERVENTIONS:
Other: anesthetics and extended information before dental treatment — The extended information is a comprehensive explanation about what to expect of the treatment and the anesthetic method, phrased in positive words and opening up for questions after information is given.
  Arms: Extended information
Other: anesthetics and standard information before dental treatment — The standard information is short and concise, telling in neutral words what to expect.
  Arms: Standard information

SUMMARY:
Information about the effectiveness of treatment has been found to reduce pain, termed placebo analgesia. In this study it will be investigated whether this finding translates to the dental clinic. It will be investigated whether information that suggested that minimal pain will be experienced during filling therapy, can reduce the pain associated with that procedure compared to a group that receives standard information. All patients will receive the same amount of anesthesia and similar procedures during filling therapy. It is predicted that extended information should reduce pain, and that the reduction in pain should be associated with a reduction in stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be treated for dental caries
* Patients should be able to read and communicate in Norwegian

Exclusion Criteria:

* Patients with life threatening diseases
* Patients taking pain killers for other reasons on the day of treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Reduction of pain | 1 hour
  Pain intensity and pain discomfort will be measured by a VAS (Visual Analog Scale). The patients will report their experience of these factors verbally, four times during the treatment session.

SECONDARY OUTCOMES:
Reduction of stress | One hour
  Stress is also measured using the VAS, i.e. using the same method as for pain. Stress or sympathetic activation is measured by using scin conductance on fingers (V-Amp (Brain Products, Munich, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Magne A Flaten, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Tannlegesenteret Madlagården, TSMG, Hafrsfjord, Norway